CLINICAL TRIAL: NCT05711953
Title: Assessment of the "PAIN LOTION" Topical Preparation for the Relief of Stiffness, Reduced Mobility, and/or Mild to Moderate Musculoskeletal or Myofascial Pain: a Prospective Pre-market, Interventional, Single Arm Investigation
Brief Title: Investigation on a Topical Cosmetic Pain Lotion (Egyfil) for Stiffness and Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contrad Swiss SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTD-SW PAIN LOTION 2021
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Pain; Muscle Rigidity
MeSH Terms: conditions — Pain; Muscle Rigidity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Egyfil Pain Lotion (Experimental): Interventional study on Egyil 50mL will be topically administered ad libitum for three days.
  Interventions: Other: Egyfil Pain Lotion

INTERVENTIONS:
Other: Egyfil Pain Lotion — Egyfil is a cosmetic product to be applied to intact skin, useful to attenuate muscolar pain and stiffness, with a novel topical formulation containing hyaluronic acid, SH-Polypeptide-6 and SH-Oligopeptide-1.
  The presence of sodium hyaluronate and peptides mixture promotes the pain alleviating activity and soothing properties of the product.

SUMMARY:
The application of a novel topical formulation for the treatment of muscular pain and stiffness (Egyfil), containing hyaluronic acid, SH-Polypeptide-6 and SH-Oligopeptide-1, is investigated to evaluate efficacy and safety in 26 patients with stiffness and pain. Single-Arm, Pre-Market, interventional study.

DETAILED DESCRIPTION:
26 male and female patients, ranging from 24 to 78 years old, will receive Egyfil Pain Lotion given for the treatment of pain and stiffness over a three-days period. The primary objective of the study is to evaluate the clinical performance of the lotion in providing relief from stiffness, reduced mobility, and muscle tension pain.

ELIGIBILITY:
Inclusion Criteria:

1. signed participants informed consent form (ICF);
2. male or Female, aged > 18 years at the time of the signature of ICF;
3. 3 to 10 rating according to the Numerical Rating Scale (NRS), applied in participants with muscle tension pain;
4. willing to follow all study procedures;
5. willing to follow indications.

Exclusion Criteria:

1. use of analgesics within the 24 hours prior to V1;
2. damaged skin in the area of treatment;
3. infective or prior inflammatory processes near the area of treatment;
4. ongoing cutaneous allergies;
5. serious and chronical pathological skin conditions (i.e., rosacea, psoriasis, vitiligo) including diagnosticated cancer with/without ongoing antitumor therapy;
6. allergy to lotion components (aqua (water), glycerin, caprylic/capric triglyceride, aloe barbadensis leaf juice powder, simmondsia chinensis seed oil (simmondsia chinensis (jojoba) seed oil), phenoxyethanol, ammonium acryloyldimethyltaurate/vp copolymer, carbomer, tocopheryl acetate, tocopherol, benzoic acid, sodium hydroxide, sodium hyaluronate, dehydroacetic acid, ethylhexylglycerin, butyrospermum parkii butter (butyrospermum parkii (shea butter)), sorbitol, SH-polypeptide 6; SH-oligopeptide-1
7. immune system illnesses;
8. uncontrolled systemic diseases;
9. known drug and/or alcohol abuse;
10. mental incapacity that precludes adequate understanding or cooperation;
11. participation in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Muscle Stiffness, measured by Numerical Rating Scale (NRS) | 3 days
  The primary efficacy endpoint of the study will be the evaluation of the clinical performance of the Egyfil, used as intended in patients affected by muscle stiffness, in terms of difference in NRS score between the end study visit and baseline visit, assessed by patients
  Minimum index score: 0. Maximum index score: 10
  0 means no stiffness
Pain, measured by Numerical Rating Scale (NRS) | 3 days
  The primary efficacy endpoint of the study will be the evaluation of the clinical performance of the Egyfil, used as intended in patients affected by Pain, in terms of difference in NRS score between the end study visit and baseline visit, assessed by patients
  Minimum index score: 0. Maximum index score: 10
  0 means no pain

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Pain Lotion when topically applied. | 3 days
  To evaluate eventual side effects of the product Egyfil through the assessment made by the Principal Investigator.
  Number of Participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Picotti, Osteopathy, Principal Investigator — Stefano Picotti - Individual Entrepeneur
Locations (1):
- Stefano Picotti, Cardano al Campo, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Picotti S, Forte L, Serrentino J. A pre-market interventional, single-arm clinical investigation of a new topical lotion based on hyaluronic acid and peptides, EGYFILTM, for the treatment of pain and stiffness in soft tissues. BMC Musculoskelet Disord. 2023 Oct 2;24(1):777. doi: 10.1186/s12891-023-06903-y. PMID 37784053